CLINICAL TRIAL: NCT00349635
Title: A Double-Blind, 3-Arm Study on Weight Loss With a Combination of Micronised Fenofibrate 267 mg and Metformin 1,700 mg Per Day Compared to Metformin 1,700 mg and to Placebo, at 6 Months, in Obese Patients, Followed by: A Double-Blind, 2-Arm Investigation of Weight-Loss Maintenance With the Same Combination of Micronised Fenofibrate 267 mg and Metformin 1,700 mg Compared to Placebo, at 6 Months, in the Responders.
Brief Title: A Controlled-Study on the Effect of a Combination of Fenofibrate and Metformin on Weight Loss and Weight Loss-Maintenance, in Obese Patients.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C LF23-0121 04 01; 2004-001731-28
Record Dates: First submitted 2006-07-06; First posted 2006-07-07 (Estimated); Last update posted 2007-09-03 (Estimated); Status verified 2007-08

CONDITIONS: Obesity
Keywords: Weight loss and diet.
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Metformin; Fenofibrate

INTERVENTIONS:
Drug: Metformin and Metformin + Fenofibrate

SUMMARY:
To investigate the effect on body weight of a combination fenofibrate and metformin on top of a moderate balanced calorie-deficit diet.

ELIGIBILITY:
Inclusion Criteria:

* Both genders, BMI ≥ 30 kg/m² and <40 kg/m².

Exclusion Criteria:

* Known abnormal thyroid hormone levels, or high thyroid stimulating hormone (TSH) level.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 148
Dates: Start 2004-10

PRIMARY OUTCOMES:
Weight

SECONDARY OUTCOMES:
Waist and hip circumference

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (3):
- Finland (3):
  - Site 1, Helsinki
  - Site 3, Kuopio
  - Site 2, Oulu